CLINICAL TRIAL: NCT06355258
Title: A Study of the Efficacy of Troxerutin in Preventing Thrombotic Events in COVID-19 Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Westlake University (Other)
Collaborators: Shaoxing Central Hospital (Other); Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20230817LX001
Record Dates: First submitted 2024-04-06; First posted 2024-04-09 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: COVID 19 Associated Coagulopathy
MeSH Terms: interventions — troxerutin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: According to the inclusion criteria, participants will be randomly divided into mild patients and severe patients, and then patients with severe disease were randomly assigned to placebo + low molecular weight heparin group or troxerutin + low molecular weight heparin group, and patients with mild disease were randomly assigned to placebo group or troxerutin group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Troxerutin+low molecular weight heparin (Experimental)
  Interventions: Drug: troxerutin + low molecular weight heparin
- Placebo+low molecular weight heparin (Placebo Comparator)
  Interventions: Drug: placebo + low molecular weight heparin
- Troxerutin (Experimental)
  Interventions: Drug: Troxerutin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Troxerutin — Oral troxerutin tablets, with a dosage of 3 tablets (60 mg/tablet) orally, twice daily
  Arms: Troxerutin
Drug: Placebo — Oral placebo tablets, with a dosage of 3 tablets (60 mg/tablet) orally, twice daily
  Arms: Placebo
Drug: placebo + low molecular weight heparin — 2000 IU LMWH once a day + Oral placebo tablets, with a dosage of 3 tablets (60 mg/tablet) orally, twice daily
  Arms: Placebo+low molecular weight heparin
Drug: troxerutin + low molecular weight heparin — 2000 IU LMWH once a day + Oral troxerutin tablets, with a dosage of 3 tablets (60 mg/tablet) orally, twice daily
  Arms: Troxerutin+low molecular weight heparin

SUMMARY:
The goal of this clinical trial is to learn if troxerutin works to prevent thrombotic events in mild or severe COVID-19 patients. It will also learn about the safety of troxerutin. The main questions it aims to answer are:

* Does troxerutin lower the number of thrombotic events in participants?
* What medical problems do participants have when taking troxerutin? Researchers will compare troxerutin to a placebo (a look-alike substance that contains no drug) to see if troxerutin works to prevent thrombotic events in COVID-19 patients.

Participants will:

* Take troxerutin or a placebo every day for 7 days.
* Visit the clinic at the first, fourth, seventh and 28th days after enrollment for checkups and tests
* Keep a diary of their symptoms and the number of times of thrombotic events, bleeding events and type II HIT-related thrombocytopenia

ELIGIBILITY:
Inclusion Criteria:

As long as the patient meets all of the following conditions, adult patients aged 18 and above are eligible for admission:

► COVID-19 patients, defined as: positive RT-PCR (upper respiratory tract or lower respiratory tract) for SARS-CoV-2.

Mild COVID-19 patients are defined as:

Symptomatic patients meeting the case definition for COVID-19 without evidence of hypoxia or pneumonia. Common symptoms include fever, cough, fatigue, anorexia, dyspnea, and myalgia. Other nonspecific symptoms include sore throat, nasal congestion, headache, diarrhea, nausea/vomiting, and loss of smell/taste.

Severe COVID-19 patients are defined as:

Adolescents or adults with clinical signs of pneumonia (i.e., fever, cough, dyspnea, tachypnea) plus one of the following:

1. Respiratory rate ≥30 breaths/min
2. Severe respiratory distress
3. Oxygen saturation (SpO₂) ≤90% in room air
4. Progressive deterioration of clinical symptoms with lung imaging showing significant progression of lesions (>50%) within 24 to 48 hours.

   * Written informed consent provided according to Chinese law (by the patient, legal guardian, or deferred consent in emergencies).

Exclusion Criteria:

Patients with any of the following conditions will be excluded from the study:

* Pregnant or lactating women.
* Postpartum (within 6 weeks).
* Extreme weight (100 kilograms).
* Clinical need for heparin therapy.
* Bleeding related to coagulation disorders, acute clinically significant bleeding, active gastrointestinal ulcers, or any organic lesions with high bleeding risk.
* Platelet count <50 x 10^9/L.
* Surgery within the last 15 days, or within 24 hours after spinal or epidural anesthesia.
* History of intracranial hemorrhage, large ischemic stroke, known intracranial malformation or tumor, acute infective endocarditis.
* Severe renal impairment (creatinine clearance <30 mL/min).
* Iodine allergy.
* Long-term use of oxygen supplementation.
* Moribund patients or those expected to die during the current hospitalization due to underlying disease.
* Patients deprived of freedom and those undergoing institutional psychiatric care.
* Ward of the state or under guardianship.
* Participation in other anticoagulant intervention studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Overall number of patients in prothrombotic state through 7 days | Through 7 days
  Assess coagulation-related parameters in patients' blood, including platelet count, prothrombin time (PT), antithrombin III activity (ATIIIa), plasma fibrinogen concentration (Fbg), and quantitative D-dimer.Patients with one or more indicators in the abnormal range, including PT < 11s (reference interval: 11-14 s), FG > 4g/L (reference interval: 2-4 g/L), D-dimer < 0.5 μg/mL (reference interval: 0-0.5 μg/mL), are considered in a prothrombotic state.

SECONDARY OUTCOMES:
Tolerability of anticoagulation therapy | Through 28 days
  Percentage of patients experiencing at least one major bleeding event (MBE) as defined by the International Society on Thrombosis and Haemostasis (ISTH) by day 28.
Adverse event | Through 28 days
  Percentage of patients experiencing at least one adverse event above grade 2

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoxing central hospital, Shaoxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided